CLINICAL TRIAL: NCT02735291
Title: Single Arm, Two Phase, Multicenter Trial to Evaluating the Efficacy and Safety of the CAR-T for Recurrent or Refractory Acute Non T Lymphocyte Leukemia
Brief Title: Study Evaluating the Efficacy and Safety With CAR-T for Recurrent or Refractory Acute Non T Lymphocyte Leukemia
Acronym: EECNTL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinobioway Cell Therapy Co., Ltd. (Industry)
Collaborators: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-06-01
Record Dates: First submitted 2016-03-29; First posted 2016-04-12 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Leukemia
Keywords: Leukemia CAR-T
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Name:The Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T) Dosage form：injection Dosage:100ml/time Frequency:The first day,the second day,29 days,injection once a day in this three days Duration:Only injection three times
  Interventions: Biological: CD19-targeted CAR-T cells

INTERVENTIONS:
Biological: CD19-targeted CAR-T cells — This study have only one arm that is CAR-T experimental arm. Firstly all participators will be attended the screening, who passed the screening for the treatment of CAR-T cells, the CAR-CD19-modified T cells can recognize and kill tumor cells in the body，follow-up 35 months..

SUMMARY:
This single-arm,multicenter Phase 2 trial will treat the patients who have recurrent or refractory acute non T lymphocyte leukemia with an infusion of the patient's own T cells that have been genetically modified to express a chimeric antigen receptor (CAR) that will bind to tumour cells that express the EPCAM protein on the cell surface.The study will determine if these modified T cells help the body's immune system eliminate tumour cells.The trial will also study the safety of treatment with CAR-T,how long CAR-T cells stay in the patient's body and the impact of this treatment on survival.

DETAILED DESCRIPTION:
This is a single-arm,multicenter Phase 2 study to evaluate the efficacy and safety of the CAR-T for recurrent or refractory acute non T lymphocyte leukemia.The study will be conducted using a phase I/II design.The study will have the following sequential phases:Part A (screening leukapheresis, cell product preparation, and cytoreductive chemotherapy) and Part B (treatment and follow-up). The follow-up period for each participant is approximately 35 months after the final CAR-T infusion. The total duration of the study is expected to be approximately 3 years. A total of 24 patients may be enrolled over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with acute non T lymphocytic leukemia after conventional treatment is invalid or recurrence of refractory, and by flow cytometry or pathological immunohistochemical examination, confirm the leukemia cells express can intervene molecular targets;
2. Age 3 to 75 years old, both male and female;
3. Is expected to survive more than 3 months;
4. Physical condition is good: 0-2 score ECOG score;
5. General requirements peripheral blood as basic normal (i.e., white blood cells >= 4.0 x10^9 / L, hemoglobin > 100 g/L, the platelet count>= 50 x10^9 / L ), progress faster, in patients with special severe fully inform the patient related risk and gain understanding and consent, peripheral blood cell index can be extended to white blood cells >= 2.0 x10^9 / L, hemoglobin > 60 g/L, the platelet count >= 30 x10^9 / L. But blood T lymphocytes in peripheral blood count must >=0.2 x10^9 / L;
6. No obvious abnormal heart, liver and kidney function (namely basic normal ecg; kidney function: Cr <=2.0 x ULN (Upper limit of normal value ); liver function: Alt/aspartate aminotransferase acuities <=2.5 x ULN, BIL<= 2.0 x ULN) , no large wounds that haven't healed on the body;
7. Into groups to participate in voluntarily, good adherence, can cooperate test observation, childbearing age women must be 7 days before starting treatment expert pregnancy test and the results were negative, and signed a written informed consent form.

Exclusion Criteria:

1. Various types of T lymphocyte leukemia, etc;
2. Organ failure, such as heart: Class III and IV; liver: to Child grading of liver function grade C; kidney: kidney failure and uremia stage; lung: symptoms of severe respiratory failure; brain: disorder of consciousness;
3. Existing serious acute infection, uncontrollable, or have fester sex and chronic infection, wound in delay no more.
4. Patients with significant graft versus host disease (GVHD) after organ transplant history or allogeneic hematopoietic stem cell transplantation;
5. Systemic autoimmune diseases or immunodeficiency disease, patients with allergic constitution.
6. Coagulation abnormalities and severe thrombosis;
7. Pregnancy and lactation women;
8. Any other chronic disease patients who have been treated with immune agents or hormone therapy;
9. Patients who have participated in other clinical trials or other clinical trials in the past 30 days
10. The Investigator believe the patients should not participate in this experiment.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The overall efficiency | 5 years
  The number of complete remission (CR) +The number of complete remission with incomplete hematologic recovery (CRi)/Total number of cases being treated

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Zhai, Professor, Principal Investigator — Chief physician; Hui Liao, Doctor, Study Director — Chief physician
Locations (2):
- China (2):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - No. 454 Hospital of People'S Liberation Army, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] An F, Wang H, Liu Z, Wu F, Zhang J, Tao Q, Li Y, Shen Y, Ruan Y, Zhang Q, Pan Y, Zhu W, Qin H, Wang Y, Fu Y, Feng Z, Zhai Z. Influence of patient characteristics on chimeric antigen receptor T cell therapy in B-cell acute lymphoblastic leukemia. Nat Commun. 2020 Nov 23;11(1):5928. doi: 10.1038/s41467-020-19774-x. PMID 33230103